CLINICAL TRIAL: NCT01319552
Title: Immunomodulatory Properties of Fresh Versus Stored Packed Red Blood Cells for Transfusion
Brief Title: Fresh Versus Old Red Blood Cells for Transfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven L. Spitalnik, Professor of Pathology, Columbia University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAAD3737; R01HL098014 (NIH)
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Iron, Abnormal Blood Level; Other Abnormal Blood Chemistry
Keywords: red blood cells; transfusion; storage; sickle cell disease; β-thalassemia; hemoglobin-associated iron
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fresh transfusion (Other): 1 unit autologous transfusion of red blood cells stored for 3-7 days under standard conditions
  Interventions: Procedure: Fresh transfusion; Procedure: Old transfusion
- Old transfusion (Experimental): 1 unit autologous transfusion of red blood cells stored for 40-42 days under standard conditions
  Interventions: Procedure: Fresh transfusion; Procedure: Old transfusion

INTERVENTIONS:
Procedure: Fresh transfusion — 1 unit autologous transfusion of red blood cells stored for 3-7 days under standard conditions
  Other Names: Stored transfusion
Procedure: Old transfusion — 1 unit autologous transfusion of red blood cells stored for 40-42 days under standard conditions
  Other Names: Stored transfusion

SUMMARY:
Packed red blood cell units destined for transfusion can be stored for up to 42 days prior to transfusion based on Food and Drug Administration (FDA) guidelines. Recent studies suggest that certain patients transfused with blood stored for longer duration have poorer outcomes than patients transfused fresher blood. The investigators' hypothesis is that the delivery of an immediate and substantial load of hemoglobin-associated iron from a stored unit of blood leads to changes that explain the differences in outcome between patients transfused old versus fresh blood. The investigators propose to test this hypothesis in humans by transfusing an individual's own blood, both fresh and after storage, and comparing levels of various outcome measures.

DETAILED DESCRIPTION:
Participants in this study will be asked to participate in a standard blood donation. The blood will be processed per standards at the investigators regional blood center (New York Blood Center) and then split into two equal units and shipped to Columbia University Medical Center for storage and transfusion. One unit will be transfused back into the same individual fresh (i.e. between 3-7 days after donation). The other unit will be transfused 42 days after donation. Blood samples will be drawn before, during, and after transfusion to measure levels of various analytes.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* male body weight >130 lbs, female body weight > 155 lbs
* male height >5'1", female height >5'5"
* hemoglobin >13.3 g/dL

Exclusion Criteria:

* ineligible for donation based on the New York Blood Center autologous blood donor questionnaire
* systolic blood pressure >180 or <90 mm Hg
* diastolic blood pressure >100 or <50 mm Hg
* heart rate <50 or >100
* temperature >99.5 F prior to donation
* temperature >100.4 F or subjective feeling of illness prior to transfusion
* positive results on standard blood donor infectious disease testing
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spitalnik L Spitalnik, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Hod EA, Brittenham GM, Billote GB, Francis RO, Ginzburg YZ, Hendrickson JE, Jhang J, Schwartz J, Sharma S, Sheth S, Sireci AN, Stephens HL, Stotler BA, Wojczyk BS, Zimring JC, Spitalnik SL. Transfusion of human volunteers with older, stored red blood cells produces extravascular hemolysis and circulating non-transferrin-bound iron. Blood. 2011 Dec 15;118(25):6675-82. doi: 10.1182/blood-2011-08-371849. Epub 2011 Oct 20. PMID 22021369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of volunteers began in December 2008 and ended in October 2010. All the volunteers were recruited at Columbia University.
Groups:
- Transfusion: Fresh transfusion : 1 unit autologous transfusion of red blood cells stored for 3-7 days under standard conditions followed by old transfusion : 1 unit autologous transfusion of red blood cells stored for 40-42 days under standard conditions
Period: Overall Study
Arm/Group | Transfusion
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Transfusion: Fresh transfusion: 1 unit autologous transfusion of red blood cells stored for 40-42 days under standard conditions
  1 unit autologous transfusion of red blood cells stored for 3-7 days under standard conditions Old transfusion: 1 unit autologous transfusion of red blood cells stored for 40-42 days under standard conditions
Arm/Group | Transfusion
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Measure of Non-transferrin-bound Iron
Description: Comparison of increase in non-transferrin-bound iron for each participant between his or her "fresh" and "old" blood transfusion four hours after transfusion.
Time Frame: four hours after transfusion
Measure: Mean (Standard Deviation); unit: μM
Groups:
- Old Transfusion: Old transfusion : 1 unit autologous transfusion of red blood cells stored for 40-42 days under standard conditions
Arm/Group | Fresh Transfusion | Old Transfusion
Number analyzed (Participants) | 14 | 14
μM | 0.16 (0.99) | 3.17 (3.26)

ADVERSE EVENTS:
Arm/Group | Transfusion
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transfusion (N=14)
Nausea (Gastrointestinal disorders) | 2 (2) — Vasovagal at time of donation
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No